CLINICAL TRIAL: NCT01536483
Title: Effects of Recto-colic Enemas of Butyrate on the Digestive Disorders of Very Low Birth Weight Preterms <1250 Grams. Clinical Trial Prospective, Monocentric, Randomized in Double-blinded.
Brief Title: Effects of Recto-colic Enemas of Butyrate on the Digestive Disorders of Very Low Birth Weight Preterms <1250 Grams
Acronym: NEOTRANS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The second intermediary analysis showed no significant difference between both arms
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRD/10/04-H
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Very Low Birth Weight Preterms
Keywords: Butyrate; Preterms; Very Low Birth Weight (<1250g); Rectocolonic enemas; Digestive maturation; Parenteral nutrition weaning; ECUN; Whole gut transit time

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Butyrate (Experimental): New born with a birth weight <1000g: Seven enemas of butyrate will be performed every 2 days from PND5
  New born with a birth weight >1000g: Seven enemas of butyrate will be performed every day from PND5
  Interventions: Drug: Butyrate enemas
- Therapeutic Abstention (No Intervention): The protocol will pretend enema: instillation in the diaper the product under consideration, to make the two indistinguishable processes (time, odor, wicking diaper ...)

INTERVENTIONS:
Drug: Butyrate enemas — Seven enemas
  * Possibility to delay from 24 to 48 hours the procedure in case of clinical poor tolerance(maximum two enemas postponed and delayed at PND12 and PND13)
  * The study remains blinded for the investigation team through the intervention of a clinical research nurse
  * According to the procedure previously described by Nakaoka et al. (2009), a lubricated Foley catheter Ch 6 will be introduced into the rectum, the balloon will be inflated with 1 ml water for injections. Butyrate solution will be placed in a bag placed 50 cm above the child. Therefore, treatment administration will be performed at a controlled pressure of 50 cm H2O without any manual intervention
  * Installation time and retention is setted at 15 minutes
  * Treatment units will be directly placed in the incubator 30 min before the procedure to warm the enema to +36°C
  * Per-treatment clinical monitoring of the tolerance will be performed by a neonatologist
  Arms: Butyrate

SUMMARY:
Clinical management of very low birth weight newborns (VLBW <1250g) consists in several challenges to adapt immature physiological systems to extrauterine life. Advances in neonatal medicine for pulmonary and/or neurological and/or cardiovascular diseases have significantly improved outcomes of these children. However, the gastro-intestinal (GI) tract remains a major cause of morbidity due to

1. the immaturity of GI functions (prolonged ileus, bacterial overgrowth and translocation),
2. the complication of GI tract immaturity: intestinal perforation and enterocolitis necrotizing)
3. the need of a prolonged parenteral nutrition and its complications (central venous catheter infections, sepsis, electrolyte disturbances) but without generate a high proof level on this targeted population (<1250g).

The GI functions are progressively acquired during development and are largely sensitive to the environment, especially the intestinal luminal content. Indeed, probiotics and prebiotics have shown beneficial effects upon GI functions of newborns. One of the metabolite of the gut flora potentially involved is the butyrate. Butyrate is a short chain fatty acid produced in the colon by the microbiota (carbo-hydrates degradation). The colonic amount of butyrate increases gradually after birth. The beneficial effects of butyrate are related to its properties upon the epithelial barrier (anti-inflammatory, antioxidant, barrier repair) and upon the enteric nervous system (network of neurons and glial cells) that regulate GI functions and in particular colonic motility.

To date, there is no clinical consensus to manage digestive disorders of VLBW. Several clinical studies have assessed the effects of prokinetic drugs, dietary supplements (probiotics, prebiotics) but without generate a high proof level on this targeted population. In this context, a recent study of our Research Unit (INSERM-CIC Mère-Enfant 004) has shown benefit effects of oral probiotics supplementation in children with birth weight greater than 1000g but not in extreme preterms with birth weight less than 1000g.

The main hypothesis to explain theses results lies in the intensive use of antibiotic and feeding interruption frequency in this targeted population which induce disturbances in the composition of the gut lumen (in particular the flora).

Colonic enemas assessed in various observational studies concerning VLBW seem to demonstrate a clinical efficiency upon the colonic transit, underlying by mechanical and osmotic mechanisms.

Here, the investigators propose to evaluate the clinical efficiency of butyrate enemas by a prospective randomized clinical trial blinded design.

The purpose of NEOTRANS study is to demonstrate that butyrate enemas may improve the nutritional management of extreme preterm less than 1250 grams, by facilitating the development of colic motility and clinical nutrition tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Any preterm infant with a birth weight less than or equal to 1250 grams admitted in the neonatal intensive care unit of Nantes Hospital
* Inborn or outborn
* No signs of gastrointestinal perforation or ECUN
* Absence of severe congenital disease
* Written informed consent of parental authority.

Exclusion Criteria:

* Newborn with birth weight greater than 1250 grams,
* Gestational age > 30 AG
* Digestive pathology diagnosed prior PND5: perforation, necrotizing enterocolitis, malformations
* Severe congenital pathology inconsistent with clinical assessment.
* Parental Refusal

Ages: 5 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2012-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of colonic butyrate enemas in digestive maturation of preterms | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  The primary outcome of NEOTRANS study consists in the evaluation of the effects of colonic butyrate enemas upon the digestive maturation of preterms.
  This endpoint is based on a clinical criteria that is the delay of weaning of the parenteral nutrition support. An increase of 25% (50 vs 75%) will be considered clinically significant.
  Parenteral nutrition weaning is defined as the day where enteral caloric intake reach 80% of total calories.

SECONDARY OUTCOMES:
Gastrointestinal complications frequency | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Nosocomial infections frequency | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Iatrogenic effect | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
whole gut transit time (red carmine test) | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Growth | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  Comparaison between 2 arms of height, weight and head circumference
Invasive ventilation support | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Bronchopulmonary dysplasia incidence | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Hospitalization duration | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
Neuromotor development | 2 years
  ASQ questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes, Nantes, France